CLINICAL TRIAL: NCT03357783
Title: Macroscopic Deciduosis in Pregnancy is Finally a Common Entity
Acronym: Deciduose
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD0315
Record Dates: First submitted 2017-11-20; First posted 2017-11-30 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Deciduitis; Complicating Pregnancy
Keywords: Frequency; Macroscopic; Deciduosis; Ovarian; Neoplasm; Pregnancy
MeSH Terms: conditions — Pregnancy Complications; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Macroscopic deciduosis — Deciduosis is a benign lesion during pregnancy that is not correlated with obstetrical complications. Our study has shown that this physiological phenomenon is more frequent that originally thought, being present in 10% of the Cesarean sections, and is associated with abdominal pain during pregnancy.

SUMMARY:
The purpose of this study is to determine the prevalence of macroscopic deciduosis found randomly in Cesarean sections and the secondary objective to determine the association with any obstetrical complications or adverse effects.

DETAILED DESCRIPTION:
Ectopic decidua or deciduosis is defined as the extrauterine location of decidual tissue and can occur in the cervix, vagina and various abdominal organs like the ovary omentum, appendix, peritoneum, the pelvic lymph nodes. Other rare sites with deciduosis include the kidneys , the lungs and even the skin . Decidualization is a physiologic process during pregnancy, under the influence of ovarian and placental steroid secretion, with total involution in the four to six week post partum period.

ELIGIBILITY:
Inclusion Criteria:

* All cesarean section

Exclusion Criteria:

* Patients refusing to participate

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All cesaren section
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2014-02-01 (Actual); Study Completion 2014-02-01 (Actual)

PRIMARY OUTCOMES:
All cases of cesarean section. | During cesarean section.
  The purpose of this study is to measure the number of participants who developed macroscopic decidosis in caesareans.

CONTACTS AND LOCATIONS:
Overall Officials: Georges MARKOU, Principal Investigator — Hôpital NOVO

IPD SHARING:
Plan to Share IPD: No